CLINICAL TRIAL: NCT04887818
Title: Assessment of Efficacy and Side Effects of Dlitiazem Ointment With Lidocaine vs. Diltiazem Ointment With Lidocaine for Treatment of Chronic Anal Fissure: Randomized Clinical Trial
Brief Title: Diltiazem Ointment With Lidocaine vs. Nifedipine Ointment With Lidocaine Ointment for Treatment of Chronic Anal Fissure
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: REB20-0239
Record Dates: First submitted 2021-04-07; First posted 2021-05-14 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-04

CONDITIONS: Fissure in Ano; Rectal Diseases; Rectal Bleed
MeSH Terms: conditions — Fissure in Ano; Rectal Diseases; Gastrointestinal Hemorrhage | interventions — Lidocaine

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial comparing efficacy and side effect profile of topical diltiazem + lidocaine vs. topical nifedipine + lidocaine
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Topical diltiazem + lidocaine (Experimental)
  Interventions: Drug: 2% Diltiazem ointment with 1.5% lidocaine
- Topical nifedipine + lidocaine (Active Comparator)
  Interventions: Drug: 0.3% Nifedipine ointment with 1.5% lidocaine

INTERVENTIONS:
Drug: 2% Diltiazem ointment with 1.5% lidocaine — 3 g of topical 2% diltiazem ointment with 1.5 % lidocaine applied in the perianal region circumferential q12h x 12 weeks
  Arms: Topical diltiazem + lidocaine
Drug: 0.3% Nifedipine ointment with 1.5% lidocaine — 3 g of topical 0.3% nifedipine ointment with 1.5 % lidocaine applied in the perianal region circumferential q12h x 12 weeks
  Arms: Topical nifedipine + lidocaine

SUMMARY:
Anal fissure is a common anorectal diseases characterized by tear of the anoderm from the dentate line to the anal verge leading to pain and bleeding during and post defecation. It may be a benign disease, but patients suffering from disease report significantly impacted quality of life especially when it becomes chronic. Several treatment modalities have been studied for chronic anal fissure, and topical calcium channel blockers (CCB) showed promising benefit and side effect profile in treatment of chronic anal fissure. Topical Diltiazem and Nifedipine are currently widely used CCBs for chronic anal fissure after multiple studies showing their benefits compared to different agents or modalities. To the investigators' knowledge, there is no study comparing the efficacy of topical Diltiazem and Nifedipine directly. The investigators aim to design a pragmatic randomized clinical trial to compare the efficacy, and side effect profile of topical Nifedipine and Diltiazem in treatment of chronic anal fissure.

DETAILED DESCRIPTION:
Anal fissure is a common anorectal diseases characterized by tear of the anoderm from the dentate line to the anal verge. It is a benign disease, but symptoms including stabbing pain during and post defecation, bleeding, and irritation lead to decreased quality of life. Acute anal fissure are superficial splits, and mostly heal spontaneously within 4 weeks with or without conservative management including high fibre diet and stool softeners. Chronic anal fissure is characterized by symptoms lasting longer than 2 months, and clinical findings of sentinel perianal skin tag, hypertrophied anal papilla, exposure of the underlying internal anal sphincter or anal cicatrization. The pathophysiology involves hypertonia of the internal anal sphincter leading to a reduction in mucosal blood flow, therefore poor healing tendency.

Several treatment modalities have been studied for chronic anal fissure. Surgical therapy (ie. lateral internal sphincterotomy) has shown promising healing rate, but its role as first line treatment was limited by significant complications including permanent flatus or fecal incontinence. Chemical sphincterotomy was introduced as a promising first line treatment due to its safe side effect profile and comparable healing rate. Topical Nitro donor initially showed a reasonable healing rate, but it was associated with high rate of significant headache leading to early termination of the therapy.

Calcium channel blockers (CCB) were then introduced to the market due to its known systemic vasodilator effect. Systemic administration of CCB is associated with various side effects including hypotension, positional hypotension, and flushing, but the topical agents were associated with minimal systemic side effects while demonstrating potent local vasodilator effect. Several randomized clinical trials have shown excellent healing rate, and safe side effect profile of both topical Diltiazem and Nifedipine. Currently, both agents are prescribed as the standard of care for first line treatment of symptomatic anal fissure.

To the investigators' knowledge, there is no study comparing the efficacy of topical Diltiazem and Nifedipine directly. The investigators aim to design a pragmatic randomized clinical trial to compare the efficacy, and side effect profile of topical Nifedipine and Diltiazem in treatment of chronic anal fissure.

This study will be a prospective, randomized, double-blinded study involving patients with chronic anal fissure undergoing 12-week treatment course of 2% Diltiazem ointment with 1.5% lidocaine vs. 0.3% Nifedipine ointment with 1.5% lidocaine. Patients with IBD, anorectal surgery, infection, radiation, instrumentation, obstetrical injuries, or patients who are currently pregnant will be excluded. Both the surgeons and the participants will be blinded from the agent being used. The participants will be followed up in the clinic at 3 months to evaluate patient reported outcome and physical exam findings of anal fissure.

Primary outcome is the anal fissure related symptoms reported by the patients upon completion of the therapy. Physical exam findings will documented and to aid in assessment of the response to the therapy, but patient reported outcome will be the most important clinical information to assess efficacy of the therapy. Secondary outcome include rate of side effects, patient compliance rate, recurrence rate, and time from cure to recurrence. Recurrence is defined by return of symptoms related to anal fissure in patients who experienced resolution of symptoms.

ELIGIBILITY:
Inclusion Criteria:

* History or clinical findings consistent with chronic anal fissure including symptoms (sharp pain during and post defecation, bleeding, or perianal irritation) with duration over 2 months
* Physical exam findings of sentinel anal skin tag, hypertrophied anal papilla, exposure of the underlying internal anal sphincter or anal cicatrization.
* Patient with history of trial of other topical agents for chronic anal fissure may be included for participation, but will be stratified based on previous treatment as they may be less likely to respond to another topical agent.
* Patient with concomitant hemorrhoids will also be included.

Exclusion Criteria:

* Patients with history of inflammatory bowel disease, perianal abscess, perianal fistula, anal cancer, anorectal instrumentation, trauma, surgery, radiation, obstetrical injuries, or current pregnancy will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Perianal pain | 12 weeks
  Perianal pain with defecation upon completion of 12-week therapy. Visual analogue pain scale will be used with 0 being no pain, and 10 being the worst pain possible.
Anal bleeding | 12 weeks
  Anal bleeding with defecation upon completion of 12-week therapy. Patient report of bleeding or no bleeding post defecation will be recorded.
Perianal irritation | 12 weeks
  Perianal irritation upon completion of 12-week therapy. Patient will report of presence of irritation or absence of irritation will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No